CLINICAL TRIAL: NCT06233357
Title: Course of Inflammation and Infection Markers in Critically Ill ICU Patients Under Casirivimab- and/or Tocilizumab Application
Brief Title: Critically Ill ICU Patients Under Casirivimab- and/or Tocilizumab Application
Acronym: CasiTocCOVID
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Principal Investigator, University of Ulm
Other Study IDs: University Ulm
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Outcome, Fatal; Tocilizumab; Interleukin 6; Critically Ill
Keywords: COVID-19; critically ill; ICU; casirivimab imdevimab; tocilizumab; interleukin 6; C-reactive protein; ferritin; procalcitonin; mortality
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — Therapeutics; imdevimab; tocilizumab; casirivimab and imdevimab drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- N, no casirivimab / imdevimab or tocilizumab: No intervention
- C, treated with casirivimab / imdevimab: Active comparator
  Interventions: Drug: treated without (N), with casirivimab / imdevimab (C) or tocilizumab (T), solely, or in combination of both (C + T)
- T, Treated with Tocilizumab: Active comparator
  Interventions: Drug: treated without (N), with casirivimab / imdevimab (C) or tocilizumab (T), solely, or in combination of both (C + T)
- C + T, treated with casirivimab / imdevimab and tocilizumab: Active comparator
  Interventions: Drug: treated without (N), with casirivimab / imdevimab (C) or tocilizumab (T), solely, or in combination of both (C + T)

INTERVENTIONS:
Drug: treated without (N), with casirivimab / imdevimab (C) or tocilizumab (T), solely, or in combination of both (C + T) — IgG seronegative SARSCoV2-Spike antibody (< 0,80 U/ml) COVID-19 patients were treated with 1 dose of subcutaneous casirivimab and imdevimab, 1200 mg (600 mg of each). Patients with CRP > 75 mg/l or IL-6 > 75 ng/l were treated with one dose of intravenous tocilizumab 8 mg/kg body weight
  Other Names: casirivimab / imdevimab; tocilizumab
  Groups: C + T, treated with casirivimab / imdevimab and tocilizumab; C, treated with casirivimab / imdevimab; T, Treated with Tocilizumab

SUMMARY:
In a retrospective observational study, critically ill COVID-19 patients admitted to the ICU with the CoV-2 delta-variant between august 2021 and february 2022 were evaluated (ethics application nr. 129/22 of the ethics commssion of the university Ulm.

DETAILED DESCRIPTION:
According to the recommendations, IgG seronegative SARSCoV2-Spike antibody (< 0,80 U/ml) COVID-19 patients were treated with 1 dose of subcutaneous casirivimab and imdevimab, 1200 mg (600 mg of each). Patients with CRP > 75 mg/l or IL-6 > 75 ng/l were treated with one dose of intravenous tocilizumab 8 mg/kg body weight. 28-day mortality and 30-day time course of leukocyte counts and serum concentrations of C-reactive protein (CRP), procalcitonin (PCT), interleukin 6 (IL-6) and ferritin in 4 patient groups, i. e., treated without (N) or with casirivimab / imdevimab (C) or tocilizumab (T), solely, or in combination of both (C + T), were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COVID-19
* CoV-2 delta-variant
* critically ill patients
* ICU

Exclusion Criteria:

* tuberculosis
* active hepatitis
* HIV

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a retrospective observational study, critically ill COVID-19 patients admitted to the ICU with the CoV-2 delta-variant between august 2021 and february 2022 were evaluated. IgG seronegative SARSCoV2-Spike antibody (< 0,80 U/ml) COVID-19 patients were treated with 1 dose of subcutaneous casirivimab and imdevimab, 1200 mg (600 mg of each). Patients with CRP > 75 mg/l or IL-6 > 75 ng/l were treated with one dose of intravenous tocilizumab 8 mg/kg body weight.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality rates in the 4 groups | 28-day mortality
  Number of survivors and nonsurvivors

SECONDARY OUTCOMES:
Leukocyte count in 4 groups | 30-days
  Routine blood analysis
C-reactive protein in 4 groups | 30-days
  Routine blood analysis over time
Interleukin 6 serum concentrations in 4 groups | 30-days
  Routine blood analysis over time
Ferritin serum concentrations in 4 groups | 30-days
  Routine blood analysis over time
Procalcitonin serum concentrations in 4 groups | 30-days
  Routine blood analysis over time

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, Principal Investigator — University of Ulm
Locations (1):
- Clinic of Anesthesiology, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No